CLINICAL TRIAL: NCT04789811
Title: The Effectiveness of Exercise and Dry Needling Treatment Combination in Patients With Nocturnal Calf Cramps
Brief Title: Exercise and Dry Needling Treatment Combination in Nocturnal Calf Cramps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kars State Hospital (Other)
Responsible Party: Principal Investigator, Fatih Bagcier, Principal Investigator, Kars State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Biruni University
Record Dates: First submitted 2021-02-27; First posted 2021-03-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Nocturnal Leg Cramps; Myofascial Pain Syndrome
Keywords: Dry needling; Calf cramp; Myofascial trigger point
MeSH Terms: conditions — Sleep-Wake Transition Disorders; Myofascial Pain Syndromes | interventions — Muscle Stretching Exercises; Dry Needling

STUDY DESIGN:
Intervention Model Description: Prospective randomised controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): It describes the exercise protocol that the patients will do.
  Interventions: Other: Stretching exercise
- Exercise plus Dry Needling Group (Experimental): It describes the exercise protocol to be performed by the patients and the methodology of dry needling to be applied.
  Interventions: Other: Stretching exercise; Other: Dry needling

INTERVENTIONS:
Other: Stretching exercise — Stretching exercise: Stretching exercises were planned for 30 seconds, ten repetitions for each stretching, 10 minutes in total, four days a week, for two weeks.
Other: Dry needling — Dry needling: A total of 3 sessions of dry needling, once a week, were applied to the gastrocnemius muscle.
  Arms: Exercise plus Dry Needling Group

SUMMARY:
The Investigators aim to evaluate the effectiveness of dry needling treatment in addition to stretching exercises on cramp duration, cramp intensity, cramp frequency, sleep quality, and sensitivity of myofascial trigger points in patients with nocturnal calf cramp.

DETAILED DESCRIPTION:
Nocturnal leg cramps are sudden, involuntary, painful contractions of the lower extremity in the nighttime, most often in the calf muscles, that gradually lessens. Its etiology is not clear. It can be seen in electrolyte disturbances, drug side effects, neuromuscular diseases, diabetes mellitus, peripheral vascular pathologies. It has been mentioned in the literature that myofascial trigger points in the gastrocnemius muscle may be associated with nocturnal calf cramps. Our aim in this study is to evaluate the effectiveness of the combination of stretching exercises and dry needling therapy on cramp duration, cramp intensity, cramp frequency, sleep quality, and algometer measurement in patients with nocturnal calf cramps and whose had myofascial trigger point in the gastrocnemius muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with only nocturnal calf cramp
* Patients with a trigger point in the unilateral gastrocnemius muscle
* Being between the ages of 18-50

Exclusion Criteria:

* Patients using diuretics or hypertension medications that may trigger cramping
* Those with a chronic disease history
* Those diagnosed with spinal stenosis
* Electrolyte disturbance in laboratory tests

Ages: 18 Years to 50 Years | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-25 (Estimated); Study Completion 2021-06-25 (Estimated)

PRIMARY OUTCOMES:
Change in calf cramp duration | 3 months
  How many seconds the patient feels cramp is questioned. Higher values represent a worse outcome
Change in Number of Cramps | 3 months
  How many times a day the patient feels cramp is recorded. Higher values represent a worse outcome
Change in cramp intensity levels with visual analog scale | 3 months
  How intense the cramp felt by the patient was recorded with a visual analog scale. The score is between 0 to 10, and higher values represent a worse outcome.
Change in algometric sensitivity measurement | 3 months
  Myofascial trigger point sensitivity in the gastrocnemius muscle was measured with an algometer. Higher scores represent a worse outcome.
Change in sleep quality | 3 months
  The sleep quality of the patients was evaluated with the Pittsburgh Sleep Quality index. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Bagcier, M.D., Principal Investigator — Kars State Hospital
Locations (1):
- Kars State Hospital, Kars, Turkey (Türkiye)